## Statistical Analysis Plan for Study Protocol: IRB-18-7223

## Role of wrist-based blood pressure monitoring in clinical practice

A pilot study to explore the feasibility and utility of around the clock wrist-based blood pressure measurements during patient transition of care

NCT03862742

October 4, 2018

## Sponsor:

Scripps Translational Science Institute (Scripps) 10550 N. Torrey Pines Road La Jolla, CA 92037

Laura Jane Nicholson, MD, PhD <a href="mailto:lnicho@scripps.edu">lnicho@scripps.edu</a>

Michael Y. Song, MD, PhD song.michael@scrippshealth.org

Steven R. Steinhubl, MD <a href="mailto:steinhub@scripps.edu">steinhub@scripps.edu</a>

Eric Topol etopol@scripps.edu

Statistical Analysis Plan (SAP): The written description of the statistical considerations for analyzing the data collected in the study. Includes how data are analyzed, what specific statistical methods are used for each analysis, and how adjustments are made for testing multiple variables. If some analysis methods require critical assumptions, the written description should allow data users to understand how those assumptions were verified.

This is a preliminary study to examine BP trends as measured by a wrist based blood pressure device. Statistical analysis will be done using two tailed student's t test, either paired or unpaired depending on the comparison, with alpha <0.05 as significance.